CLINICAL TRIAL: NCT03148041
Title: The Effectiveness of Health Education Program on Level of Awareness of Stroke Among Population at Risk Attending Primary Health Care Center, Jeddah, Saudi Arabia, a Randomized Control Field Trial
Brief Title: The Effect of Health Education Program on Level of Awareness for Stroke Among Population
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Taibah University (Other)
Responsible Party: Principal Investigator, ibrahim rashad noor elahi, Principle investigator Dr Ibrahim Rashad Noor Elahi, MD, MPH, Taibah University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: Dr Ibrahim Rashad Noor Elahi
Record Dates: First submitted 2017-05-05; First posted 2017-05-10 (Actual); Last update posted 2017-10-19 (Actual); Status verified 2017-10

CONDITIONS: Stroke
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- intensive health education program (Active Comparator): Participants in the intervention group will have an intensive health education program of the introductory lecture and brochures about stroke as well as they fill up the questionnaire at baseline. At week 6 and 12 of the study the participants will only fill up the questionnaire.
  Interventions: Other: health education program
- routine care (Placebo Comparator): Participants in the control group will have a routine care of different lecture and brochures than the intervention group as well as they fill up the questionnaire at baseline. At week 6 and 12 of the study the participants will only fill up the questionnaire.
  Interventions: Other: health education program

INTERVENTIONS:
Other: health education program — Intensive health education program for intervention group: 1.The introductory 30 minute Arabic lecture for increase level of the awareness of the participants regarding stroke. Lecture from the USA National Stroke Association, 2011, will be used. The lecture includes the following issues about stroke (1) definition; (2) signs and symptoms; (3) risk factors; (4) treatment; and (5) prevention.
  2. Self-help materials will involve health education brochures regarding stroke and will be distributed for all participants at the time they are attending the lecture. The brochures which will be used for this study will be collected from the World Stroke Day 2016 Brochures, the Arabic version.
  The routine care for control group: different lecture and brochures will be used

SUMMARY:
The investigator of this study would like to test the hypothesis of the effectiveness of health education program on level of awareness of stroke among population at risk whom attending the primary health care center in Jeddah, in Saudi Arabia. The investigator will divide the participants into two groups. The intervention group whom will have the intensive health education program, and the control group whom will have the routine care. Participants will be followed up for 3 months to assess the effect of different health education programs on their level of awareness about stroke. Also The investigator will relate different socioeconomic factors to level of awareness.

DETAILED DESCRIPTION:
The aim of the current study is to increase level of the awareness regarding risk factors and warning signs of stroke among population at risk who attending the primary health care center at Jeddah city in Saudi Arabia.

The primary objective of this study is to assess the effectiveness of the health education program on the level of the awareness and knowledge gain among population at risk attending primary health care center, Jeddah, Saudi Arabia.

The secondary objective of this study is to relate the effect the socioeconomic factors of the participants on the level of the knowledge and the awareness regarding stroke.

The current study will be conducted at primary health care center (PHCC) at Jeddah city of the western province of Saudi Arabia. Within Jeddah city, there are 46 PHCCs. In this research, The investigator will select one PHCC to be included in this study. Selection of the PHCC will be based on the simple random technique. Letter to the public health administration for permission to be included in this study will be prepared by the principle investigator of this study and will be sent before conducting this study.

This study adopted an open-label, randomized control field trial design. Participants who are registered and followed up in the primary health care center will be included in this study. The eligibility criteria for the participants included in this study involved both male and female of 40 year old or more of different body weights, and able to speak Arabic. Participants with at least one risk factor like hypertensive, diabetic, and dyslipidemia will be included in this study. A family member of any participants will be excluded and will not participate in this study.

The number of participants required will be 45 people for each the intervention and the control group (α=0.05, β=0.8).

In this research, The investigator will select one PHCC by simple random technique. Once a center agrees to participate, signs a covenant of agreement and identifies a center champion.

Participants will be recruited from the PHCC congregation. Recruitment for participants will take about 1 month of duration. The process of recruitment will be held at the physicians' clinics and will be conducted by the principle investigator of this study.

A trained nurse will help in the recruitment process. After meeting the participants in the clinic, the next step will be checking the eligibility criteria and baseline data collection of the participants. After checking the eligibility for the participants, The investigator will ask them whether they would like to participate in this study or not. If the participants are willing to participate, they will signed the informed consent for this study. After that,The investigator will make a phone call and text a message to the participants' mobile phone to invite them to participate in this study. The phones' numbers of the participants will be collected from their files.

After recruitment of the participants, The investigator will conduct a stratified block randomization method. Stratification will be based upon age groups and gender. Age groups involve participants from age 40 -50 year, 51-60 year, and those above 60 year of age. Participants will also stratified to male and female. The total number of strata for this study will be 6 strata.

Randomization will be performed within each stratum, and it will be blocked. Within each block, participants will be randomized, by simple random method, to receive either the intervention group (will receive intensive health education program), or to the control group (will receive the routine care). Hence there are two different treatment group (intervention, and control), the block size is of minimum of four. To avoid selection bias of the participants, The investigator will use different random block sizes from 6-12.

Although contamination is not a major issue in this study, The investigator will try to keep the intervention and the control group of the participants apart from each other to eliminate threats to internal validity through interactions between the participants. A family member of any participants will be excluded and will not participate in this study.

For better controlling for those who might be lost during the study's period, the percentage of those participants LTFU will be calculated, whether or not they are equal for the intervention and the control group, and whether those LTFU have different baseline characteristics and prognosis than those who completed the study. Also, the investigator will make frequent contacts (at least twice) with all participants upon recruitment to insure not to lose any of them, and in case of lose any of them, the investigator will clarify the reasons for that. Later, in the analysis of this study, the investigator will apply an interim analysis and will use the worst-case scenario and will apply the intention to treat (ITT) analysis.

The eligible participants of this study will be recruited in the intervention group or in the control group through randomization as mentioned above. Participants in an intervention group will receive an intensive health education program for 3 months. In comparison, participants in the control group will receive a routine care for the same period of time. The principle investigator of this study will assure to give both programs to the intervention and to the control group.

Both primary and secondary outcomes data of this study will be collected at baseline, at 6 weeks, and at 12 week of follow-up for both the intervention and the control group. At baseline, participants in the intervention group will receive an introductory lecture about stroke and a self-help materials, and they will fill up the questionnaire. Participants in the control group will have different lecture and brochures, as well as they will fill up the same questionnaire delivered to the intervention group.

The introductory lecture about stroke will comprise of 30 minute Arabic lecture that will be developed to increase level of the awareness of the participants regarding stroke. Here, a lecture from the USA National Stroke Association, 2011, will be used. Translation and validation of this lecture will be done by the principle investigator of this study. The lecture includes the following issues: (1) definition of stroke; (2) signs and symptoms of stroke; (3) risk factors of stroke; (4) treatment of stroke; and (5) prevention of stroke. The lecture will be available to all participants upon requested. Here, a permission from the author to give this lecture will be assured, as well as three expert panel will be involved; two neurologists' expert opinion, and one community medicine specialist opinion.

Self-help materials will involve health education brochures regarding stroke and will be distributed for all participants at the time they are attending the lecture. The brochures which will be used for this study will be collected from the World Stroke Day 2016 Brochures, the Arabic version.

At baseline, at 6 weeks, and at 12 week of follow up, all participants will fill up an interview questionnaire identified by the American Heart Association. This questionnaire consists of items pertaining to warning symptoms of stroke and heart attack (HA) as well as cardiovascular diseases (CVD). The structured questionnaire contained 18 items, including 9 items for stroke and 9 items for HA warn¬ing symptoms, as well as 11 items for CVD risk factors.

For this study, the items for stroke and those related to the awareness of stroke risk factors will be included in the questionnaire. One point will be given for each correct answer and a zero will be given for each incorrect answer; then individual scores will be added to obtain a total score.

In addition, the participants will also be asked what they would do if they thought someone was having a stroke, and their ability to perceive the possible occurrence of a stroke will assessed. This questionnaire will be completed by all participants and will be supervised by the study's principle investigator before and immediately after attending the introductory lecture of the stroke.

The questionnaire will be translated into Arabic, approved, and be checked for its content validity by the expert panel of this study. Then the questionnaire will be tested for both comprehension and readability during a pilot study on 10 participants whom will be not included in the final analysis of the entire study. The questionnaire include the following components: gender, age group, education level, monthly income, and knowledge of stroke risk factors. Besides that, marital status, employment status, obesity, smoking and its duration, hypertension, diabetic, and dyslipidemia diseases and their duration, and area of residency (rural/urban) will be added to this questionnaire as they are important risk factors that might be related to stroke.

Accurate response rates of stroke symptoms by the participants in 9 items will include: sudden dizziness, sudden numbness or weakness of the arm or leg, especially on one side of the body, sudden trouble speaking or understanding, sudden trouble walking, loss of balance or coordination, sudden numbness or weakness of the face especially on one side of the body, sudden confusion, sudden severe headache with no known cause, sudden trouble seeing in one or both eyes, and nausea or vomiting.

In this study, the investigator will attempt to make frequent contact (at least twice) with the participants in the control group to limit the possibility that a difference between treatment groups in outcome is due to greater attention paid to the intervention group.

Physical activities, dietary pattern, smoking status, cardiac disorders (atrial fibrillation, valvular heart disease, myocardial infarction, coronary artery disease, congestive heart failure, and electrocardiographic evidence of left ventricular hypertrophy), and family history of stroke among first-degree relatives, will be recorded in this study.

ELIGIBILITY:
Inclusion Criteria:

* The eligibility criteria for the participants included in this study involved both male and female of 40 year old or more of different body weights, and able to speak Arabic. Participants with at least one risk factor like hypertensive, diabetic, and dyslipidemia will be included in this study.

Exclusion Criteria:

* A family member of any participants will be excluded and will not participate in this study.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2017-11-01 (Estimated); Primary Completion 2017-12-30 (Estimated); Study Completion 2018-03-02 (Estimated)

PRIMARY OUTCOMES:
Calculate the score level of awareness of stroke symptoms | The outcome 1 will be assessed at baseline, 6 weeks, and 12 week of study.
  Accurate response rates of stroke symptoms that included in the questionnaire. It will be scored out of 9.

SECONDARY OUTCOMES:
Calculate the percentage of the socioeconomics factors that identified by the participants as risk factors for stroke. | The outcome 2 will be assessed at baseline, 6 weeks, and 12 week of study.
  Different socioeconomic risk factors of stroke will be identified by the participants during filling up the questionnaire.Then the percentage of those factors will be calculated by the study investigator.

CONTACTS AND LOCATIONS:
Overall Officials: farah A mansuri, professor, Study Chair — Taibah University

IPD SHARING:
Plan to Share IPD: Undecided